CLINICAL TRIAL: NCT07383246
Title: 68Ga-CTR-FAPI PET-CT-guided Precision Surgery for Newly Diagnosed Medullary Thyroid Carcinoma: A Multicenter, Open-labeled, Randomized Controlled Phase 3 Trial
Brief Title: CTR-FAPI-guided Precision Surgery for Newly Diagnosed MTC
Acronym: CAST-MTC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Peking Union Medical College Hospital (Other); Peking University Cancer Hospital & Institute (Other); Peking University First Hospital (Other); Xiangya Hospital of Central South University (Other); Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other)
Responsible Party: Principal Investigator, SHAOYAN LIU, Director of Head and Neck Surgery, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAST-MTC-01
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Medullary Thyroid Carcinoma
Keywords: Medullary Thyroid Cariconma; Surgery; CTR-FAPI
MeSH Terms: conditions — Carcinoma, Medullary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ⁶⁸Ga-CTR-FAPI PET-CT guided surgery (Experimental): The participants assigned to the experimental arm will undergo ⁶⁸Ga-CTR-FAPI PET-CT imaging.
  The surgical extent will be determined by ⁶⁸Ga-CTR-FAPI PET-CT image.
  Interventions: Procedure: 68Ga-CTR-FAPI PET-CT guided surgery
- investigator choice of surgery (Active Comparator): Since there is currently no standardized surgical extent for medullary thyroid carcinoma, the surgical approach for the control group will be determined by the attending surgeon, based on routine preoperative evaluation.
  Interventions: Procedure: investigator choice of surgery

INTERVENTIONS:
Procedure: 68Ga-CTR-FAPI PET-CT guided surgery — The participant will be intravenously administered with [68Ga]Ga-CTR-FAPI and undergo PET-CT imaging.The surgical extent will be determined by [68Ga]Ga-CTR-FAPI PET-CT image. The minimum extent of resection is total thyroidectomy plus central neck dissection. Therapeutic dissection of the lateral neck compartment and upper mediastinal lymph nodes within standard boundaries is performed, with the extent determined based on CTR-FAPI findings.
  Arms: ⁶⁸Ga-CTR-FAPI PET-CT guided surgery
Procedure: investigator choice of surgery — Since there is currently no standardized surgical extent for medullary thyroid carcinoma, the surgical approach for the control group will be determined by the attending surgeon. Including but not limited to: Surgery based on conventional imaging (ultrasound/CT); Prophylactic neck dissection; Surgery based on tumor size, germline RET mutation status, and state of central lymph node metastasis; Surgery based on intraoperative frozen section findings.
  Arms: investigator choice of surgery

SUMMARY:
This is a multicenter, randomized, open-label, non-inferiority Phase III clinical trial, aims to compare 68Ga-CTR-FAPI PET-CT-guided surgery to investigator-chosen surgical approaches to evaluate its efficacy in treating newly diagnosed medullary thyroid carcinoma. This study plans to enroll 150 newly diagnosed MTC patients, who will be randomly assigned in a 2:1 ratio to the experimental group (surgery based on 68Ga-CTR-FAPI PET-CT findings) and the control group (surgery based on the investigator's choice). The primary endpoint is the biochemical cure rate, with secondary endpoints including the biochemical cure rate in the R0 resection subgroup, the unnecessary dissection rate in the biochemical-cured subgroup, 3-year recurrence-free survival, the rate of change in surgical extent, and diagnostic accuracy.

DETAILED DESCRIPTION:
Medullary thyroid carcinoma (MTC) is a relatively difficult-to-treat malignant thyroid tumor with a wide range of metastases. Surgery is the only curative treatment, and accurate assessment of the extent of metastatic disease is crucial for planning the surgical extent. Conventional imaging modalities have limited utility in fully evaluating the extent of MTC involvement. The tumor microenvironment of MTC is rich in cancer-associated fibroblasts (CAFs), which highly express fibroblast activation protein (FAP), whereas normal tissue fibroblasts express little to no FAP. Given the co-localization relationship between MTC cells and CAFs, fibroblast activation protein inhibitors (FAPIs) targeting FAP can be used to localize MTC lesions. The molecular probe CTR-FAPI, developed through covalent modification, improved the detection rate and diagnostic accuracy for MTC, providing a theoretical basis for performing precise surgery for MTC based on the extent of disease revealed by 68Ga-CTR-FAPI PET-CT.

This is a multicenter, randomized, open-label, two-arm, non-inferiority Phase III clinical trial. This study plans to enroll 150 newly diagnosed MTC patients, who will be randomly assigned in a 2:1 ratio to the experimental group (surgery based on 68Ga-CTR-FAPI PET-CT findings) and the control group (surgery based on the investigator's choice).

The study hypothesizes that CTR-FAPI-guided surgery can identify and resect more positive lesions while avoiding prophylactic dissection of disease-free areas, thereby benefiting patients. Proving the benefit of the former requires complete resection of all positive lesions. However, due to the frequent local invasion and adhesions associated with MTC lesions, achieving R0 resection is difficult in some patients. Therefore, the primary objective is to demonstrate that CTR-FAPI-guided surgery is non-inferior to the investigator's choice in IIT population. The primary endpoint was biochemical cure rate at 1-month post-surgery, defined by normalization of serum calcitonin levels. This parameter represents the strictest curative level for MTC and correlates with survival outcomes. In a nationwide retrospective analysis involving 863 patients, the 10-year overall survival (OS) of biochemical-cured MTC was 97.7%; in comparison, the 10-year OS of non-cured MTC was 70.3%.

The secondary objectives are to demonstrate its superiority in the subgroup achieving R0 resection, and to show that it avoids unnecessary lateral neck/upper mediastinum dissection in the subgroup achieving biochemical-cure. Key secondary endpoints include: the biochemical cure rate at 1 month post-surgery in the R0 resection subgroup, and the unnecessary dissection rate in the biochemical-cured subgroup, which address the two important secondary objectives and the study hypothesis. Other secondary endpoints include: 3-year recurrence-free survival, the rate of surgical plan modification in the experimental group, and the diagnostic accuracy of different imaging modalities for MTC lesions.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed medullary thyroid carcinoma meeting either criterion a or criteria b + c:

  1. Pathologically or cytologically confirmed diagnosis;
  2. Elevated serum calcitonin level (>10 pg/mL);
  3. Other infectious or neoplastic diseases excluded.
* Life expectancy ≥ 12 weeks;
* ECOG performance status of 0 or 1;
* Absence of distant metastasis confirmed by conventional imaging, with resectable locoregional disease;
* Scheduled to undergo surgery within 30 days;
* Females of childbearing potential must use effective contraception (e.g., sterilization, intrauterine device, condoms, oral/injectable contraceptives, abstinence, or partner vasectomy) during the study and for 6 months after study completion. Male participants must agree to use effective contraception during the same period;
* Capable of understanding and voluntarily signing the informed consent form with good compliance.

Exclusion Criteria:

* History of prior treatment for medullary thyroid carcinoma (e.g., surgery, radiotherapy, targeted therapy, radionuclide therapy, or interventional therapy).
* Major organ dysfunction, defined as:

  1. Bone marrow impairment: WBC ≤ 4.0×10⁹/L or neutrophils ≤ 1.5×10⁹/L; platelets ≤ 100×10⁹/L; hemoglobin ≤ 90 g/L
  2. Hepatic impairment: PT or APTT ≥ 1.5 × ULN; total bilirubin ≥ 1.5 × ULN; ALT/AST ≥ 2.5 × ULN (or ≥ 5 × ULN in participants with liver metastases); ALP ≥ 2.5 × ULN (or ≥ 4.5 × ULN in cases with bone or liver metastases)
  3. Renal impairment: BUN ≥ 1.5 × ULN; serum creatinine ≥ 1.5 × ULN
* Women who are planning pregnancy, currently pregnant, or breastfeeding.
* History of other malignant tumors;
* Inability to lie flat for at least 30 minutes;
* Known allergy to contrast agents;
* Claustrophobia or other psychiatric disorders that may preclude compliance with study procedures;
* Unwillingness to participate in the clinical trial;
* Assessed as not being a surgical candidate or refusal to undergo surgery;
* Any other condition deemed by the investigator to make the participant unsuitable for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical cure rate | 1 month after surgery
  Biochemical cure is defined as postoperative serum calcitonin level less than 10pg/ml

SECONDARY OUTCOMES:
Biochemical cure rate in R0 resection subgroup | 1 month after surgery
  Biochemical cure is defined as postoperative serum calcitonin level less than 10pg/ml. The outcome is assessed in the R0 resecton subgroup.
Unnecessary dissection rate in the biochemical cured subgroup | 1month after surgery (after pathogoly report issued)
  The unnecessary dissection rate is defined as the proportion of patients whose dissections outside the central compartment yield no metastatic lymph nodes. This outcome will be evaluated exclusively in the biochemically cured subgroup, as only surgeries that achieve biochemical cure are considered to have an adequate surgical extent. In these patients, any dissection that yields negative specimens is deemed unnecessary. We anticipate that CTR-FAPI imaging will enable precise surgical planning, allowing for a more reduced extent of dissection compared to prophylactic surgery, thus minimizing complications.
Recurrence-free survival | 3 years after surgery
  Recurrence-free survival is defined as the peroid from the date of surgery until any recurrence revealed by structural imaging or any cause of death. The day of imaging examination will be regarded as the day of recurrence.
Change rate in the extent of surgery in the experimental arm | immedaite after surgery
  Change rate in the extent of surgery compared to the investigator's chioce in the experimental arm. The investigator's chosen surgical extent will be documented preoperatively when the attending doctor is not exposed to the CTR-FAPI findings.
Diagnostic accuracy rate | 1 month after surgery (after pathology report issued)
  Diagnostic accuracy is defined as the proportion of correctly diagnosed lesions (including both positive and negative) to the total number of lesions documented. It will be calculated separately for different imaging modalities (CTR-FAPI PET-CT, ultrasound, and CT).

CONTACTS AND LOCATIONS:
Overall Officials: Shaoyan Liu, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kong Z, Li Z, Cui XY, Wang J, Xu M, Liu Y, Chen J, Ni S, Zhang Z, Fan X, Huang J, Lin Y, Sun Y, He Y, Lin X, Meng T, Li H, Song Y, Peng B, An C, Gao C, Li N, Liu C, Zhu Y, Yang Z, Liu Z, Liu S. CTR-FAPI PET Enables Precision Management of Medullary Thyroid Carcinoma. Cancer Discov. 2025 Feb 7;15(2):316-328. doi: 10.1158/2159-8290.CD-24-0897. PMID 39470165
- [Result] Cui XY, Li Z, Kong Z, Liu Y, Meng H, Wen Z, Wang C, Chen J, Xu M, Li Y, Gao J, Zhu W, Hao Z, Huo L, Liu S, Yang Z, Liu Z. Covalent targeted radioligands potentiate radionuclide therapy. Nature. 2024 Jun;630(8015):206-213. doi: 10.1038/s41586-024-07461-6. Epub 2024 May 22. PMID 38778111